CLINICAL TRIAL: NCT04699825
Title: Cardiovascular Changes in the Infants of Mothers With Preeclampsia and Factors Associated With Neonatal Outcomes
Brief Title: Cardiovascular Changes in Infants of Preeclampsia Mother
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ASAli, Assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: cardiovascularpreeclampsia
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Circulation

STUDY DESIGN:
Intervention Model Description: enrollment of infants born from preeclampsia mother and control from infants born from normal pregnancies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): new-born infants born from preeclampsia mother
  Interventions: Other: Cardiovascular and immunological changes
- control group (Other): new-born infants born from mothers with normal pregnancy matched with the same gestational age, sex and race
  Interventions: Other: Cardiovascular and immunological changes

INTERVENTIONS:
Other: Cardiovascular and immunological changes — performing cardiac ultrasound, vascular doppler, and immunological study on cord blood sample

SUMMARY:
Preeclampsia (hypertension during pregnancy) is a common problem affecting 2-8% of pregnancies worldwide and is typically diagnosed by increased blood pressure and proteinuria. The rate of preeclampsia has increased since the 1980s with higher rates at extreme maternal ages as well as during the first pregnancy. Pre-eclampsia is a serious hypertensive disorder of pregnancy affecting outcomes for both mother and infants. These infants not only have increased risk of neonatal complications including preterm birth, intrauterine growth restriction, abnormal Doppler parameters, feed intolerance, intestinal problem, poor growth, and long term lung condition but also have increased risk of cerebral palsy, abnormal neurodevelopmental outcomes, cardiovascular disease, stroke, and mental disorders during childhood and adulthood.

DETAILED DESCRIPTION:
Preeclampsia is diagnosed according to the International Society for the Study of Hypertension in Pregnancy (ISSHP) criteria: BP > 140/90 on two occasions in previous normotensive mother after 20 weeks of gestation and one of the following; proteinuria in urine > 0.3 gram/kg/day or acute kidney or liver dysfunction or signs of uterine dysfunction. The onset of preeclampsia can be early before 34 weeks of pregnancy (Early-onset preeclampsia) or late after 34 weeks of pregnancy (Late-onset preeclampsia). Early-onset preeclampsia, especially between 28-32 weeks gestation, is characterized by a high prevalence of microvascular changes in the placenta that makes mothers and their infants are more liable to complication. The pathogenesis of preeclampsia is unclear.

Preeclampsia affects hematopoiesis and the fetal myeloid lineage leading to thrombocytopenia, neutropenia, decrease phagocytic function, decrease T regulatory cells, and an increase in cytotoxic natural killer cells in neonates. Innate and adaptive immunity are regulated by myeloid cells and the immune changes in infants of preeclampsia mothers could lead to increased incidence of neonatal sepsis and the development of chronic inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Infants born from Pregnant women with preeclampsia, their mother willing to give consent.

Exclusion Criteria:

* 1-Infant with a major heart problem.
* Infants with major congenital and genetic anomalies.

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac changes | within 72 hours after birth
  cardiac output will be presented by ml/minute
Cardiac function changes | within 72 hours after birth
  Fractional shortening and ejection fraction will be presented by percentage
Vascular changes in superior mesenteric and anterior cerebral arteries | 72 hours after birth
  Doppler parameters( peak-systolic velocity, end-diastolic velocity, and mean velocity.
  All will be measured in meter/second

SECONDARY OUTCOMES:
Feeding problem | 3 months after birth
  rate of necrotizing enterocolitis and feeding intolerance
oval all outcomes | 3 months
  Rate of long term lung condition, sepsis, intraventricular hemorrhage and overall mortality
immunological changes | cord blood at birth
  interleukins level

IPD SHARING:
Plan to Share IPD: No
No, we will take consent from participant in this study only.

REFERENCES:
- [Background] Ananth CV, Keyes KM, Wapner RJ. Pre-eclampsia rates in the United States, 1980-2010: age-period-cohort analysis. BMJ. 2013 Nov 7;347:f6564. doi: 10.1136/bmj.f6564. PMID 24201165
- [Background] Hansen AR, Barnes CM, Folkman J, McElrath TF. Maternal preeclampsia predicts the development of bronchopulmonary dysplasia. J Pediatr. 2010 Apr;156(4):532-6. doi: 10.1016/j.jpeds.2009.10.018. Epub 2009 Dec 14. PMID 20004912
- [Background] Marins LR, Anizelli LB, Romanowski MD, Sarquis AL. How does preeclampsia affect neonates? Highlights in the disease's immunity. J Matern Fetal Neonatal Med. 2019 Apr;32(7):1205-1212. doi: 10.1080/14767058.2017.1401996. Epub 2017 Nov 20. PMID 29113524
- [Background] Bujold E, Chaiworapongsa T, Romero R, Gervasi MT, Espinoza J, Goncalves LF, Berman S, Yoon BH, Kim YM. Neonates born to pre-eclamptic mothers have a higher percentage of natural killer cells (CD3-/CD56+16+) in umbilical cord blood than those without pre-eclampsia. J Matern Fetal Neonatal Med. 2003 Nov;14(5):305-12. doi: 10.1080/jmf.14.5.305.312. PMID 14986803
- [Background] Ness RB, Sibai BM. Shared and disparate components of the pathophysiologies of fetal growth restriction and preeclampsia. Am J Obstet Gynecol. 2006 Jul;195(1):40-9. doi: 10.1016/j.ajog.2005.07.049. Epub 2006 Apr 21. PMID 16813742